CLINICAL TRIAL: NCT05039190
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Seamless and Group Sequential Phase 2/3 Study to Evaluate the Efficacy and Safety of HBM9161 (HL161) Subcutaneous Injection in Patients With Generalized Myasthenia Gravis
Brief Title: Evaluate the Efficacy and Safety of HBM9161(HL161)Subcutaneous Injection in Patients With Generalized MG Patients
Acronym: MG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9161.3 ph3
Record Dates: First submitted 2021-08-29; First posted 2021-09-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Myasthenia Gravis
Keywords: MG
MeSH Terms: conditions — Myasthenia Gravis | interventions — HBM9161

STUDY DESIGN:
Intervention Model Description: To confirm the efficacy of HBM9161 subcutaneous injection for the treatment of gMG in Chinese patientsTreatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: HBM9161 (680mg ) (Active Comparator): HBM9161 680mg; First treatment period: Subcutaneous injection, QW for 6 doses; Second treatment period: Subcutaneous injection, QW for 6 doses
  Interventions: Drug: HBM9161 Injection (680mg)
- Placebo Comparator: Placebo (Placebo Comparator): Placebo; First treatment period: Subcutaneous injection, QW for 6 doses; Second treatment period: Subcutaneous injection, QW for 6 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9161 Injection (680mg) — HBM9161 Injection
  Arms: Experimental: HBM9161 (680mg )
Drug: Placebo — Placebo Injection
  Arms: Placebo Comparator: Placebo

SUMMARY:
Primary study objective: To confirm the efficacy of HBM9161 subcutaneous injection for the treatment of gMG in Chinese patients

DETAILED DESCRIPTION:
This is the phase 3 part of a multi-center, randomized, double-blind, placebo-controlled, group sequential designed, seamless phase 2/3 study to confirm the efficacy and safety of HBM9161 (HL161) subcutaneous injection for the treatment of gMG in patients with generalized myasthenia gravis.

Study drug will be administrated by cycle. Each cycle consists of 5-week treatment period, followed by a 4-week observation period (9 weeks in total). During the 5-week treatment period, subjects will receive 6 doses of study drug (HBM9161 680 mg or matching placebo) by subcutaneous injection, once a week (QW). After the 5-week treatment period, subjects will be followed up weekly to assess efficacy and safety. After the completion of first treatment cycle, subjects may start the second cycle of treatment if re-treatment criteria are met. Otherwise, subjects will be followed up weekly until they are eligible for the second cycle or the end of the study, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form (ICF).
2. Male or female ≥ 18 years of age at the screening visit.
3. Female subjects must meet the following conditions to participate in this study:

   1. Not of childbearing potential (ie, physiologically incapable of becoming pregnant, including women who have been postmenopausal for 2 or more years);
   2. Of potential childbearing potential, have a negative serum pregnancy test result at the screening visit, and agree to adhere to one of the following acceptable effective methods of contraception (ie, per approved product label insert and physician instructions) consistently and correctly during the study, until 60 days after the last dose:

   i. Total abstinence (based on subject preference and previous lifestyle); or ii. Implantation of a levonorgestrel implant at least 1 month prior to study drug administration, but no longer than 3 years; or iii. Injection of a progestogen at least 1 month prior to study drug administration; or iv. A cycle of oral contraceptives (combined contraceptives or progestin-only) for at least 1 month prior to study drug administration; or v. Double contraception: condom or cervical cap (diaphragm or cervical cap) plus spermicide (foam/gel/cream/suppository); or vi. An intrauterine device, implanted by a qualified physician; or vii. Estrogen vaginal ring; or viii. Contraceptive patch.
4. Male subjects must use effective contraceptive methods or have their heterosexual partners use effective contraceptive methods during their participation in this clinical trial.
5. Meets MGFA myasthenia gravis clinical classification IIa-IVa (includes types IIa, IIb, IIIa, IIIb, and IVa) at the screening visit and at the baseline visit.
6. Screening and baseline MG-ADL score ≥ 5, and < 50% of them is from ocular muscle.At least one stable background MG treatment at randomization.Positive or negative AchR-Ab/MUSK-Ab at the screening visit and meets at least 1 of the following 3 criteria:

   1. Repeated electrical stimulation indicates neuromuscular junction transmission disorder (including medical history record);
   2. Positive Tensilon test or neostigmine test (including medical history record);
   3. The patient's MG symptoms improve after treatment with oral cholinesterase inhibitors at the judge of the physician.
7. Results from clinical laboratory tests at screening must be acceptable to the investigator.

Exclusion Criteria:

1. Has a serious illness or condition other than myasthenia gravis that, in the judgment of the investigator, would put the subject at risk because of participation in the study, or that would affect the results of the study and the subject's ability to participate in the study.
2. Females who are pregnant or lactating or planning to become pregnant during the study period, or females of childbearing potential who are not using an effective method of contraception.
3. Subjects with severe myasthenia gravis (such as Type IVb or V) who are judged by the investigator to be inappropriate for this study (e.g., expected to require artificial assisted ventilation during the study).
4. Thymectomy performed < 12 months prior to screening.
5. Presence of other autoimmune diseases (such as uncontrolled thyroid disease, severe rheumatoid arthritis, etc.) that may affect the efficacy assessment of the study drug or affect participation in this study.
6. Has received a vaccine injection (including the COVID-19 vaccine) 4 weeks prior to the Screening Visit or is scheduled to receive a vaccine injection during the study.
7. Any active infection at the Screening Visit or serious infection requiring treatment with intravenous anti-infective drugs or hospitalization within 8 weeks before the Screening Visit.
8. Current or past 1 year alcohol or drug dependence/abuse, except nicotine and coffee.
9. Subjects who are allergic to the trial drug or its components; or history of clinically significant allergic disease (including drug allergies, anaphylaxis) that, in the opinion of the investigator, affects the subject's participation in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
In the first treatment cycle, percentage of patients with sustained improvement based on Myasthenia Gravis Activities of Daily Living Scale (MG-ADL), among serum AChR-Ab- or MuSK-Ab-positive subjects | baseline to Day 64
  Definition of sustained improvement based on MG-ADL: during the treatment cycle (5-week treatment period plus 4-week observation period), a reduction of ≥ 3 points from the baseline of MG-ADL score for 4 consecutive weekly MG-ADL assessments

SECONDARY OUTCOMES:
In the first treatment cycle, percentage of patients with sustained improvement based on MG-ADL, among all study subjects, regardless of , regardless of AChR-Ab and MuSK-Ab serologic status | Baseline to Day 64
In the first treatment cycle, percentage of subjects with sustained improvement based on Quantitative Myasthenia Gravis Scale (QMG), among serum AChR-Ab- or MuSK-Ab-positive subjects [ Time Frame: baseline to Day 64 ] | Baseline to Day 64
  Definition of sustained improvement based on QMG: a reduction of ≥ 3 points from the baseline of QMG score for 4 consecutive weekly QMG assessments during the treatment cycle (5-week treatment period plus 4-week observation period)
During the 24-study period, the proportion of weekly MG-ADL assessments that are improved ≥ 3 points from baseline among serum AChR-Ab- or MuSK-Ab-positive subjects | baseline to Day 64
In the first treatment cycle, percentage of serum AChR-Ab- or MuSK-Ab-positive subjects who meet the minimal symptom manifestation (MSE, defined as MG-ADL being 0 or 1) criterion at any visit | baseline to Day 64
Within the first 2 weeks of the first treatment cycle, percentage of AChR-Ab- or MuSK-Ab-positive subjects whose MG-ADL improved by ≥3 points from baseline | baseline to Day 64
Within the second treatment cycle, percentage of patients with sustained improvement based on MG-ADL, among serum AChR-Ab- or MuSK-Ab-positive subjects during the second 9-week treatment cycle | baseline to Day 64

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yan C, Yue Y, Guan Y, Bu B, Ke Q, Duan R, Deng H, Xue Q, Jiang H, Xiao F, Yang H, Chang T, Zou Z, Li H, Tan S, Xiao H, Zhou H, Zhang H, Meng Q, Li W, Li W, Guo J, Zhang Y, Li Z, Tu J, Shi J, Li W, Lee M, Chen Y, Tao X, Zhao S, Li P, Zhao C; Batoclimab Study Team. Batoclimab vs Placebo for Generalized Myasthenia Gravis: A Randomized Clinical Trial. JAMA Neurol. 2024 Mar 4;81(4):336-45. doi: 10.1001/jamaneurol.2024.0044. Online ahead of print. PMID 38436998

DOCUMENTS (1):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT05039190/Prot_000.pdf